CLINICAL TRIAL: NCT07082036
Title: Study of the Stability of Post-stroke Hemiparetic Patients During a Task Involving Picking up an Object on the Ground. Reflection Questioning the Conventional Rehabilitation of These Patients
Brief Title: Stability of Hemiparetic Patients During a Daily Complex Task
Acronym: HemiSym
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230812; 2024-A00043-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-05-21; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hemiparesis
Keywords: Hemiparetic patients; Stability; Orientation; Postural control; Strategy; Motion
MeSH Terms: conditions — Paresis; Orientation, Spatial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Among the repercussions of hemiparesis following stroke, disturbed stability is responsible for a high risk of falls. Picking up objects from the ground, frequently trained in rehabilitation due to its risk of falling and its frequency in daily life, is a task requiring balance. To date, however, it has been little studied. We suggest that stability conditions the asymmetry adopted by patients. We hypothesise that asymmetric support at the expense of the paretic lower limb provides better stability during an unstable functional task (picking up an object from the ground) compared with the symmetrical support traditionally imposed in rehabilitation.

Postural control involves stability (maintaining balance despite constraints) and orientation (posture adopted, such as the distribution of supports). Hemiparetic patients show a lack of stability and, with regard to orientation, an asymmetry in the distribution of body weight to the detriment of the paretic limb. Symmetrisation of weight distribution has been one of the predominant concepts in rehabilitation.

DETAILED DESCRIPTION:
To analyse the stability of hemiparetic stroke patients when picking up an object on the ground in a spontaneous condition compared with a condition of imposed support symmetry.

To analyse and compare the stability, spontaneous symmetry and duration of picking up the object in a complex situation (distant target) compared with the near target in stroke patients and healthy subjects.

To explore strategy and performance of picking up the object regarding clinical outcomes (falls, sensori-motor impairments, balance..) To compare strategy of patients with right and left stroke.

ELIGIBILITY:
Inclusion Criteria:

All:

Male or female ≥ 18 years

For patients :

* Haemiparesis after a single unilateral hemispheric Stroke.
* Stroke ≥ 6 months
* Asymmetry of support between the 2 lower limbs (distribution of body weight) in a standing position at the expense of the paretic lower limb > 10%.
* Able to stand alone, without technical aids or equipment, with feet the width of the pelvis
* Able to pick up an object from the ground alone (minimum score 3/4 item 9 of the Berg Balance Scale).
* Patient informed and having signed a consent form

For healthy subjects:

- Similar characteristics (in terms of sex, age range and BMI class) to those of one of the patients already included.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemiparetic patients following stroke; Healthy subjects (same age, height, weight).
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
stability parameter: the range of the medio-lateral centre of pressure during the object picking up task | at baseline
  Two forceplate platforms. 3 trials for each condition

SECONDARY OUTCOMES:
Velocity of the centre of pressure | at baseline
  Mean velocity and in each place, in mm/s, obtained with forceplat plateforms under feet of participants during the object picking up task.
Ellipse area of the centre of pressure | at baseline
  With 95% confidence, in mm², obtained with forceplat plateforms under feet of participants during the object picking up task
Range of the centre of pressure | at baseline
  Range in antero-posterior plane, in mm, obtained with forceplat plateforms during the object picking up task
Percentage of weight bearing | at baseline
  Under each lower limb, in %, obtained with forceplat plateforms during the object picking up task
Kinematics parameters | at baseline
  range of movements of trunk, pelvis and lower limbs (hip, knee, ankle), in degrees, obtained with the optoelectronic system during the object picking up task
Questionnaires : Confidence perception and stability perception during the object picking up task | at baseline
  On a visual scale 0 (no confidence) to 10 (perfect confidence)
Clinical scales - Berg balance scale | at baseline
Clinical scales-Medical Research Council | at baseline
Clinical scales-Modified Ashworth | at baseline
Clinical scales-Nottingham Sensory Assessment | at baseline
Clinical scales -Neglect and lateropulsion scale | at baseline
Cognitive scale : Batterie Rapide d'Efficience Frontale | at baseline
Activities-Specific Balance Confidence | at baseline
Functional reach test | at baseline
  In cm

CONTACTS AND LOCATIONS:
Overall Officials: Céline Bonnyaud, Principal Investigator — Motion Analysis Laboratory, CHU Raymond Poincaré - APHP
Locations (1):
- CHU Raymond Poincaré - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided